CLINICAL TRIAL: NCT06445647
Title: Effect of Core Stability Exercise Training on Activities of Daily Living, Fatigue Level and Balance in Hemodialysis
Brief Title: Effect of Core Exercise on ADL in Hemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Lecturer of Physical therapy, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: core exercise
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis
Keywords: Core Exercise; ADL; Balance; Hemodialysis
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Active Comparator): 30 hemodialysis patient
  Interventions: Other: core Stability exercise; Other: Breathing exercises
- Control group (Active Comparator): 30 hemodialysis patient
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: core Stability exercise — core stability exercise training
  Arms: Study Group
Other: Breathing exercises — Deep breathing and diaphragmatic breathing exercises

SUMMARY:
Finding the effect of core stability exercises with breathing exercises on Activities of daily living (ADLs), fatigue level and balance in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
Sixty patients will be randomly assigned into two equal groups, the experimental (EX) group and the control group (CON). The participants' age will be 50-65 years and undergo hemodialysis. The Ex-group will attend three sessions/week of core stability exercise training (CSE) combined with Deep Breathing (25:30-min) for 8 weeks, the CON will attend 3 sessions/week of Deep Breathing (15-min) for 8 weeks. All the patients received only routine hemodialysis department care.

ELIGIBILITY:
Inclusion Criteria:

* Adults ranging from 55- 70 years old of both genders.
* Diagnosed as maintenance hemodialysis for at least 6 months or more.
* Free from mental illness, neuromuscular disorders, and serious lung problems and able to implement the interventional exercise.

Exclusion Criteria:

* Obesity (BMI ≥ 30 kg/m2)
* Orthopeadics or neurological problems that interferes with training.
* History of pulmonary problems (COPD, pneumonia)
* History of Myocardial infarction and/or cardiothoracic surgery
* Unstable medical status
* Dementia that interferes with the ability to follow instructions.
* History Chronic Fatigue Syndrome (CFS).

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Livings (ADLs) | up to 8 weeks
  ADLs will be assessed by Barthel Index (BI)
Fatigue | up to 8 weeks
  Fatigue will be assessed by fatigue assessment scale. The total score ranges from 10 to 50. A total score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Balance | up to 8 weeks
  Balance will be assessed by berg balance scale, the balance score ranges from 0 to 56, with lower scores indicating increased risk of balance loss and higher scores indicating improved functional mobility. Time up and go test (TUG)n Score < 10 seconds = normal < 20 seconds = good mobility; can walk outside alone; does not require a walking aid < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Saif, Principal Investigator — National institute for Gerontology
Locations (1):
- Kz hospital, Cairo, Egypt